CLINICAL TRIAL: NCT00874510
Title: Interventions to Improve Fatigue Management Among Physician Trainees
Brief Title: A Randomized Controlled Trial of Mandatory Naps for Physicians in Training
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EDU 08-429
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Fatigue
Keywords: sleep deprivation; fatigue
MeSH Terms: conditions — Fatigue; Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Schedule (No Intervention): interns work standard schedule, being on duty for 30 continuous hours
- Mandatory Naps (Experimental): interns on overnight extended duty shifts have mandatory sign out of cell phones and cross-coverage responsibilities for 5 hours roughly between 12 and 5 am. For Year 2, this will be two 3 hour shifts, the first between 12am-3am and the 2nd between 3am-6am.
  Interventions: Behavioral: Mandatory Naps

INTERVENTIONS:
Behavioral: Mandatory Naps — As above, interns on extended duty overnight call shifts will be required to transfer cell phones and cross-coverage responsibilities to night float residents for a 5 hour period each night they are on call. For Year 2, interns will nap in shifts, instead of concurrently, with the first nap shift between 12am-3am and the second shift between 3am-6am
  Arms: Mandatory Naps

SUMMARY:
This study will consist of a randomized controlled trial in which the investigators test the feasibility and effectiveness of mandatory nap programs for physicians in training. One site will be the general medical service of the Philadelphia Veterans Affairs Medical Center. The other will be the oncology service of the Hospital of the University of Pennsylvania. The primary outcome will be the amount slept while on call. The first year will test the efficacy of a 5 hour mandatory nap schedule, the second year will test the efficacy of a 3 hour mandatory nap schedule.

DETAILED DESCRIPTION:
Background: The release of the Institute of Medicine report on resident work hours and patient safety highlighted the risks to patient and resident safety of extended duty on-call shifts.

Objectives: The purpose of this study is to test the feasibility and effectiveness of mandatory naps during extended duty overnight shifts for residents.

Methods: For each site (PVAMC and HUP), every other month residents will be randomized to either work the standard schedule (which involves interns being on duty for 30 continuous hours) vs. the mandatory nap schedule, which involves interns signing out their beepers for 5 hours in the middle of the night to covering night floats and for 3 hours in Year 2. The primary outcome will be the amount slept as measured by actigraphs, with secondary outcomes of cognitive alertness measured by 3-minute psychomotor vigilance testing (PVT), Stanford sleepiness Scale, and other measures of resident and patient well-being.

Status: Recruitment complete, analyses phase only

ELIGIBILITY:
Inclusion Criteria:

* Residents in the University of Pennsylvania Internal Medicine Training Program who are rotating through either Philadelphia VA Medical Center Medical Service or Hospital of University of Pennsylvania Oncology Service

Exclusion Criteria:

* Refusal to consent to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G. Volpp, MD PhD, Principal Investigator — VA Medical Center, Philadelphia
Locations (1):
- VA Medical Center, Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Volpp KG, Shea JA, Small DS, Basner M, Zhu J, Norton L, Ecker A, Novak C, Bellini LM, Dine CJ, Mollicone DJ, Dinges DF. Effect of a protected sleep period on hours slept during extended overnight in-hospital duty hours among medical interns: a randomized trial. JAMA. 2012 Dec 5;308(21):2208-17. doi: 10.1001/jama.2012.34490. PMID 23212498
- [Result] Halpern SD, Kohn R, Dornbrand-Lo A, Metkus T, Asch DA, Volpp KG. Lottery-based versus fixed incentives to increase clinicians' response to surveys. Health Serv Res. 2011 Oct;46(5):1663-74. doi: 10.1111/j.1475-6773.2011.01264.x. Epub 2011 Apr 14. PMID 21492159
- [Result] Shea JA, Dinges DF, Small DS, Basner M, Zhu J, Norton L, Ecker AJ, Novak C, Bellini LM, Dine CJ, Mollicone DJ, Volpp KG. A randomized trial of a three-hour protected nap period in a medicine training program: sleep, alertness, and patient outcomes. Acad Med. 2014 Mar;89(3):452-9. doi: 10.1097/ACM.0000000000000144. PMID 24448046
- [Derived] Basner M, Dinges DF, Shea JA, Small DS, Zhu J, Norton L, Ecker AJ, Novak C, Bellini LM, Volpp KG. Sleep and Alertness in Medical Interns and Residents: An Observational Study on the Role of Extended Shifts. Sleep. 2017 Apr 1;40(4):zsx027. doi: 10.1093/sleep/zsx027. PMID 28329124

RESULTS

PARTICIPANT FLOW:
Period: Year 1
Arm/Group | Standard Schedule | Mandatory Naps
Started | 88 | 85
Completed | 88 | 85
Not Completed | 0 | 0
Period: Year 2
Arm/Group | Standard Schedule | Mandatory Naps
Started | 92 | 87
Completed | 92 | 87
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Characteristics of control and intervention groups comprised of medicine interns participating in a randomized trial of a Year 1 5-hour and Year 2 3-hour protected nap period at the Philadelphia Veterans Administration Medical Center ( PVAMC) and the Hospital of the University of Pennsylvania
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Schedule | Mandatory Naps | Total
Number analyzed (Participants) | 180 | 172 | 352
Age, Customized [Mean (Standard Deviation); unit: years]
  Year 1 PVAMC | 27.5 (2.3) | 27.3 (2.3) | 27.4 (2.3)
  Year 1 HUP | 28.1 (2.2) | 27.7 (2.0) | 27.9 (2.1)
  Year 2 PVAMC | 27.9 (2.4) | 27.9 (3.5) | 27.9 (2.9)
  Year 2 HUP | 28.1 (2.9) | 28.3 (3.0) | 28.2 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 85 | 178
  Male | 87 | 87 | 174
Region of Enrollment [Number; unit: participants]
  United States | 180 | 172 | 352

OUTCOME MEASURES:

1. Primary Outcome: Hours Slept on Overnight Extended Duty Call Shifts
Description: Two sites were separately analyzed for Mean Sleep Time for both Year 1 and Year 2.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: hours
Units Other Than Participants: Days studied
Groups:
- Arm 1 - Standard Schedule for Years 1 and Year 2: interns work standard schedule, being on duty for 30 continuous hours
- Arm 2 - Mandatory Nap: In Year 1 interns on overnight extended duty shifts have mandatory sign out of cell phones and cross-coverage responsibilities for 5 hours roughly between 12 and 5 am and were asked to nap during this time
  For Year 2, the mandatory sign out of cell phones and cross-coverage responsibilities was split between two 3 hour shifts, the first between 12am-3am and the 2nd between 3am-6am and were asked to nap during this time
Arm/Group | Arm 1 - Standard Schedule for Years 1 and Year 2 | Arm 2 - Mandatory Nap
Number analyzed (Participants) | 180 | 172
Number analyzed (Days studied) | 4159 | 4354
hours
  Sleep time Year 1 PVAMC | 1.98 [1.68 to 2.28] | 2.86 [2.57 to 3.10]
  Sleep time Year 1 HUP | 2.04 [1.79 to 2.24] | 3.04 [2.77 to 3.45]
  Sleep time Year 2 early shift PVAMC | 1.90 [1.71 to 2.10] | 2.33 [2.07 to 2.58]
  Sleep time Year 2 late shift PVAMC | 1.90 [1.71 to 2.10] | 2.40 [2.12 to 2.69]
  Sleep time Year 2 early shift HUP | 1.55 [1.36 to 1.73] | 2.40 [2.12 to 2.67]
  Sleep time Year 2 late shift HUP | 1.55 [1.36 to 1.73] | 2.44 [2.17 to 2.71]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from time of first shift of intern or resident through the end of the year study period.
Groups:
- Arm 1 - Standard Schedule: interns work standard schedule, being on duty for 30 continuous hours
- Arm 2 - Mandatory Naps: interns on overnight extended duty shifts have mandatory sign out of cell phones and cross-coverage responsibilities for 5 hours roughly between 12 and 5 am. For Year 2, this will be two 3 hour shifts, the first between 12am-3am and the 2nd between 3am-6am.
  Mandatory Naps: As above, interns on extended duty overnight call shifts will be required to transfer cell phones and cross-coverage responsibilities to night float residents for a 5 hour period each night they are on call. For Year 2, interns will nap in shifts, instead of concurrently, with the first nap shift between 12am-3am and the second shift between 3am-6am
Arm/Group | Arm 1 - Standard Schedule | Arm 2 - Mandatory Naps
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/172
Other Adverse Events (participants affected / at risk) | 0/180 | 0/172

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No